CLINICAL TRIAL: NCT06055426
Title: The Effect of Bed Bath Applied to Palliative Care Patients on Saturation, Pain Level and Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Sevil PAMUK CEBECİ, Asst.Prof.Dr., Eskisehir Osmangazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-4
Record Dates: First submitted 2023-09-11; First posted 2023-09-26 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Palliative Care
Keywords: Palliative care; nursing care; pain; sleep quality; bed bath; saturation level
MeSH Terms: conditions — Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bed bath (Experimental): Bed bath application stages:
  * Environmental elements (ambient temperature, airflow and curtain-screen) are taken under control in the clinic (Ensure that the ambient temperature is 23-24℃).
  Interventions: Other: bed bath application

INTERVENTIONS:
Other: bed bath application — Patients who agree to participate in the research and are assigned to the experimental group will receive a bed bath. In order to examine the short-term, medium-term and long-term effects of bed bath, it is planned to have the whole body bed bath performed by the researcher nurse xx three times a week, two days apart.

SUMMARY:
The research showed that bed bath applied to palliative care patients in Eskişehir City Hospital Palliative Care Service; It was planned as a randomized experimental study with a pretest-posttest control group design to determine its effect on saturation, pain level and sleep quality.

DETAILED DESCRIPTION:
Considering the individual's comfort and stabilization of vital signs, bathing practice, which is one of the independent roles of nursing; It should be applied with the right method at healthy intervals. Considering the studies on bathing in bed or in the shower; It has been observed that bathing increases patients' oxygen saturation, ensures effective breathing, reduces blood pressure and body temperature, ensures skin integrity, increases patient comfort and quality of life, and reduces anxiety levels (Uğur, 2018). In their study, Downey and Lloyd (2008) emphasize that bed bathing in hospitalized patients is important for personal cleanliness, well-being and preventing the development of infection. According to this study report, the improvement of communication between the nurse and the individual provides nurses with the opportunity to evaluate the daily activities of patient individuals. The nurse evaluates the patients' independence or dependency in activities such as individual hygiene, mobility, excretion and clothing, and thus obtains information about the individual's nutrition, sleep patterns and whether he or she has pain. It is also stated that such communication allows the individual to express his/her opinions about care, treatment or daily practices. In Erçin's (2006) study, in which the effect of early and late period bed bathing on mixed venous oxygen saturation after coronary artery bypass graft application was evaluated, no difference was seen between the control and experimental groups, while it was determined that the mixed venous oxygen saturation of both groups increased during bed bathing.

In the literature; The number of studies on the effects of bed bath application on palliative care patient groups, who frequently experience sleep disturbance and pain, is quite limited. With this study, it is aimed to contribute to the literature.

The universe of the research; It consists of patients hospitalized in the Palliative Care Clinics of a hospital in Eskişehir, Turkey. The sample size was calculated with the G power program based on the effect size obtained from the literature. The observed effect size for the parameters to be measured between groups was calculated as 0.95. According to these results, according to the power analysis calculated with 95% power and 0.05 significance level based on the two-way hypothesis in the experimental and control groups, it was calculated that a total of 60 individuals should participate in the study, at least 21 in the experimental group and 21 in the control group. This analysis was calculated with the G Power program version 3.1.

Research hypotheses

H1: Bed bath applied to palliative care patients has the effect of increasing the saturation level of the patients.

H2: Bed bath applied to palliative care patients has an effect on reducing the pain level of the patients.

H3: Bed bath applied to palliative care patients has an effect on improving the sleep quality of patients.

Randomization Method: Participants will be assigned to the experimental and control groups using the simple randomization method. Patients will be given a number starting from 1 according to the order of admission.

Patients who accepted to participate in the study and were assigned to the experimental group will be given a bed bath. In order to examine the short-term, medium-term and long-term effects of the bath, it is planned to have a whole body bed bath performed by researcher nurse XX three times a week, two days apart.

* Richard-Campbell Sleep Scale, Wong-Baker Facial Pain Scale will be applied and oxygen saturation will be measured before and after bed bath.
* The control group patients will not be given a bed bath, their measurements will be made simultaneously with the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* The first degree relative who voluntarily accepted to participate in the research gave consent to participate in the research,
* 18 years and older,
* Receiving inpatient treatment and care in the palliative care service,
* Patients who do not have bed bath application restrictions will be included.

Exclusion Criteria:

* Those who do not voluntarily agree to participate in the research,
* Under 18 years of age,
* Not receiving inpatient treatment and care in the palliative care service,
* Patients who are restricted from using bed baths will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
H1: Bed bath applied to palliative care patients has a saturation regulating effect | 1 weeks
  A form was prepared by the researcher. Partial oxygen saturation levels of the patients before, during and after the bath will be measured with the devices (pulse oximeter) used in the clinic where the research will be conducted and recorded on this form.
H3: Bed bath applied to palliative care patients has an effect on the patients' sleep quality. | 1 weeks
  The scale developed by Richards in 1987; It is a scale consisting of 6 items that evaluates the depth of night sleep, the time it takes to fall asleep, the frequency of waking up, the time spent awake when waking up, the quality of sleep and the noise level in the environment. The validity and reliability of the scale in our country was conducted by Karaman Özlü and Özer in 2015. It will be measured using the Richard-Campbell Sleep Scale. The scale consists of 6 items that evaluate the depth of night sleep, the time it takes to fall asleep, the frequency of waking up, the time spent awake when waking up, the quality of sleep and the noise level in the environment. It is evaluated on a chart between 0 and 100 using the visual analog scale technique. A score between "0-25" from the scale indicates very poor sleep, and a score between "76-100" indicates very good sleep.quality of patients.
H2: Bed bath applied to palliative care patients has an effect on changing the pain level of the patients. | 1 weeks
  Pain will be measured with the Wong-Baker Facial Pain Scale. It was developed by Wong and Baker in 1988. It is a practical and valid measurement tool for the evaluation of cancer-related pain. Patients' pain levels are evaluated by counting their facial expressions. In this scoring, which is done by numbering facial expressions, as the number value increases, the facial expression changes, which indicates an increase in the level of pain.
  0-No pain, 2-The pain is very little, 4-The pain is a little more, 6-The pain is even greater, 8-The pain is quite intense, 10-pain means the worst level of pain (Wong and Baker, 1988).

CONTACTS AND LOCATIONS:
Overall Officials: Mihraç Topçu, Principal Investigator — mihrac.topcu1@gmail.com
Locations (1):
- Sevil PAMUK CEBECİ, Eskişehir, Odunpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No